CLINICAL TRIAL: NCT06141707
Title: Adaptation and Validation of Pediatric Sleep Questionnaire (PSQ) in Arabic
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Wafaa Helmy Abdelhakeem, Principal Investigator, Minia University
Other Study IDs: Arabic Validation of PSQ
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea, pediatric sleep questionnaire
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OSA group: This group will include 66 parents in charge of participants with SRBDs.
  Interventions: Other: Arabic pediatric sleep questionnaire
- reliability group: To test the reliability of the Arabic Pediatric Sleep Questionnaire (APSQ); 33 parents in charge will be randomly selected among the 66 parents in charge of subjects with SRBDs in OSA group.
  Interventions: Other: Arabic pediatric sleep questionnaire
- control group: control group will include 66 children with no OSA
  Interventions: Other: Arabic pediatric sleep questionnaire

INTERVENTIONS:
Other: Arabic pediatric sleep questionnaire — Pediatric Sleep Questionnaire (PSQ) developed and validated by chervil et al. (2000) is a 22 item questionnaire which had been shown to have a sensitivity of 81% and specificity of 87% for SRBD.These scales for childhood SRBDs, snoring, sleepiness, and behavior are valid and reliable instruments that can be used to identify SRBDs or associated symptom-constructs in clinical research when polysomnography is not feasible.

SUMMARY:
The gold-standard in the diagnosis of Sleep-Related Breathing Disorders (SRBDs) is polysomnography, but the time, effort, and expense of laboratory studies has limited relevant research and particularly epidemiological research that requires large samples. Research in adults has profited from the existence of several validated questionnaire instruments to assess for Sleep-Related Breathing Disorders (SRBDs) or related symptoms. Pediatric Sleep Questionnaire (PSQ) developed and validated by chervil et al. (2000) is a 22 item questionnaire which had been shown to have a sensitivity of 81% and specificity of 87% for SRBDs.

In this study 152 parents in charge of children and adolescents with and without SRBDs aged from 2 years to 18 years, will participate. collection of the study sample will take place in Phoniatric clinic and otolaryngology clinic, minna University Hospital. This sample will be divided into three groups: G1, G2, and G3.

The validation of the Arabic Pediatric Sleep Questionnaire (APSQ) will be executed in many stages:

1. Translation, linguistic and cultural adaptation with bilingual Phoniatrician and qualified translator who will perform translation and back translation.
2. Pilot study with the application of the translated version on a group of SRBDs participants "20 children and adolescents with SRBDs ".
3. History will be taken from all groups.
4. Application of the survey in its final version on participants with and without SRBDs.

DETAILED DESCRIPTION:
The gold-standard in the diagnosis of Sleep-Related Breathing Disorders (SRBDs) is polysomnography, but the time, effort, and expense of laboratory studies has limited relevant research and particularly epidemiological research that requires large samples. Research in adults has profited from the existence of several validated questionnaire instruments to assess for SRBDs or related symptoms .

Pediatric Sleep Questionnaire (PSQ) developed and validated by chervil et al. (2000) is a 22 item questionnaire which had been shown to have a sensitivity of 81% and specificity of 87% for SRBDs.

This study aims at performing the validation of the Arabic version of the Pediatric Sleep Questionnaire (PSQ), called Arabic Pediatric Sleep Questionnaire (APSQ) by means of translation and cultural adaptation of the instrument and by obtaining psychometric measures of validity and reliability, to verify if the presence of childhood SRBDs and prominent symptom complexes, including snoring, daytime sleepiness, and related behavioral disturbances and to obtain normal scores for pediatric population as regard the APSQ.

In this study 152 parents in charge of children and adolescents with and without SRBDs aged from 2 years to 18 years, will participate. collection of the study sample will take place in Phoniatric clinic and otolaryngology clinic, minna University Hospital. This sample will be divided into three groups: G1, G2, and G3.

The validation of the Arabic Pediatric Sleep Questionnaire (APSQ) will be executed in many stages:

1. Translation, linguistic and cultural adaptation with bilingual Phoniatrician and qualified translator who will perform translation and back translation.
2. Pilot study with the application of the translated version on a group of SRBDs participants "20 children and adolescents with SRBDs ".
3. History will be taken from all groups.
4. Application of the survey in its final version on participants with and without SRBDs.

ELIGIBILITY:
Inclusion Criteria:

* children with obstructive sleep apnea.
* Age is from 2 to 18 years.

Exclusion Criteria:

* Presence of acute infection in the upper airway.
* Previous treatment.
* Previously diagnosed neurological or psychiatric disorder

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children diagnosed as obstructive sleep apnea
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
total score | baseline
  total score in degree

CONTACTS AND LOCATIONS:
Overall Officials: Fatma W Shahin, MD, Study Director — Minia University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chervin RD, Hedger K, Dillon JE, Pituch KJ. Pediatric sleep questionnaire (PSQ): validity and reliability of scales for sleep-disordered breathing, snoring, sleepiness, and behavioral problems. Sleep Med. 2000 Feb 1;1(1):21-32. doi: 10.1016/s1389-9457(99)00009-x. PMID 10733617